CLINICAL TRIAL: NCT01831414
Title: Etude Pilote évaluant l'Effet du Niveau d'Immersion Sur la Fonction Respiratoire Des Patients tétraplégiques bénéficiant de balnéothérapie
Brief Title: Effect of Immersion Level on Respiratory Function of Spinal Cord Injury Patients During Balneotherapy
Acronym: BALNEORESPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2009-A00246-51
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Spinal Cord Injury
Keywords: Lung function; Water immersion; Balneotherapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water immersion at cervical level (Experimental): Lung function of spinal cord injury patients will be studied with a water immersion at cervical level
  Interventions: Other: Water immersion at cervical level
- Water immersion at xyphoid level (Experimental): Lung volumes of spinal cord injury patients will be studied with a Water immersion at xyphoid level
  Interventions: Other: Water immersion at xyphoid level

INTERVENTIONS:
Other: Water immersion at cervical level — balneotherapy session of spinal cord patients with a Water immersion at cervical level
  Arms: Water immersion at cervical level
Other: Water immersion at xyphoid level — balneotherapy session of spinal cord patients with a Water immersion at xyphoid level
  Arms: Water immersion at xyphoid level

SUMMARY:
Balneotherapy is a physiotherapy technique which allows patients to work out in a weightless environment and which is often used in patients with spinal cord injury. In normal subjects, water immersion generates a reduction in lung volumes. The effects of water immersion on the respiratory function of spinal cord injury patient (who are liable to present a respiratory failure secondary to paralysis) are not well known. They could be deleterious (by majoring respiratory failure)or beneficial (by mimicking the effect of a corset and improving respiratory function). Therefore, we are planning to study the effect of different water immersion levels on the respiratory function of spinal cord injury patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient
* complete tetraplegia from spinal cord injury
* initial spinal cord injury at leat 3 months before study

Exclusion Criteria:

* contra indication to a balneotherapy session (bed-sore, skin infection or irritation, urinary or fecal incontinency, tracheostomy, ongoing infection)
* unstable respiratory state (patient free of respiratory infection or encumbrance)
* refusal to participate to the protocol
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Lung volumes | 1 hour
  Measurement of lung volumes (Vital capacity, Forced Expiratory volume at 1 second and total lung capacity) measured by standard pulmonary function test

SECONDARY OUTCOMES:
Respiratory comfort | 1 hour
  Respiratory comfort is evaluated with a visual analogical scale (ranked from 0 to 10) and the Borg dyspnea score

CONTACTS AND LOCATIONS:
Overall Officials: HELENE PRIGENT, MDPHD, Principal Investigator — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France